CLINICAL TRIAL: NCT02600819
Title: A Phase 3b Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of E/C/F/TAF Fixed Dose Combination (FDC) in HIV-1 Infected Subjects on Chronic Hemodialysis
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of E/C/F/TAF Fixed Dose Combination (FDC) in HIV-1 Infected Adults on Chronic Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-1825; 2015-002713-30 (EudraCT Number)
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: HIV-1 Infection
Keywords: End stage renal disease; Hemodialysis; Open-label; HIV-1 Infection
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E/C/F/TAF (Experimental): Participants will switch their current antiretroviral regimen to E/C/F/TAF and receive treatment for 96 weeks. After Week 96, participants in the United States (US) who wish to participate in the open-label (OL) rollover extension will continue to take E/C/F/TAF FDC until the End of E/C/F/TAF Visit.
  Interventions: Drug: E/C/F/TAF
- Open-Label Rollover Extension B/F/TAF (Experimental): At Week 96 or the End of E/C/F/TAF Visit (whichever occurs last), participants will be given the option to receive open-label bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) for at least 48 weeks.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablets administered orally once daily
  Other Names: Genvoya®
  Arms: E/C/F/TAF
Drug: B/F/TAF — 50/200/25 mg FDC tablets administered orally once daily
  Other Names: Biktarvy®
  Arms: Open-Label Rollover Extension B/F/TAF

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) fixed-dose combination (FDC) in human immunodeficiency virus (HIV-1) infected adults with end-stage renal disease (ESRD) on chronic hemodialysis (HD).

ELIGIBILITY:
Key Inclusion Criteria:

* Currently on a stable antiretroviral regimen for ≥ 6 consecutive months
* Plasma HIV-1 ribonucleic acid (RNA) concentrations < 50 copies/mL for ≥ 6 months preceding the screening visit and have HIV-1 RNA < 50 copies/mL at screening
* No documented history of HIV-1 resistance to elvitegravir (EVG), emtricitabine (FTC), lamivudine (3TC) or tenofovir (TFV) and no history of switching off EVG, FTC, 3TC or TFV due to concern for resistance
* Cluster determinant 4 (CD4+) T cell count ≥ 200 cells/μL
* ESRD with estimated glomerular filtration rate (eGFR) < 15 mL/min by Cockcroft-Gault formula for creatinine clearance
* On chronic HD for ≥ 6 months prior to screening
* Adequate hematologic function (absolute neutrophil count ≥ 1,000/mm^3; platelets ≥ 50,000/mm^3; hemoglobin ≥ 8.5 g/dL)

Key Exclusion Criteria:

* Hepatitis B co-infection
* Any clinical history, condition, or test result that, in the opinion of the Investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements
* Administration of other investigational agents (unless approved by Gilead Sciences). Participation in any other clinical trial, including observational trials, without prior approval from the sponsor is prohibited while participating in this trial.
* History or presence of allergy or intolerance to the study drugs or their components
* A new acquired immunodeficiency syndrome (AIDS)-defining condition (excluding CD4+ T cell count and percentage criteria) diagnosed within the 30 days prior to screening, with the exception of oropharyngeal candidiasis
* Received solid organ or bone marrow transplant

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (26):
- United States (19):
  - Peter J Ruane MD Inc, Los Angeles, California
  - University of California Davis, Sacramento, California
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - Infectious Disease Consultants, M.D., P.A. d/b/a Orlando Immunology Center, Orlando, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - The Research Institute, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Prime Health Care Services - St Michael's LLC d/b/a Saint Michael's Medical Center, Newark, New Jersey
  - University of North Carolina at Chapel Hill / UNC School of Medicine, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Med Center, Cincinnati, Ohio
  - MetroHealth Medical Center IRB, Cleveland, Ohio
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Trinity Health and Wellness Center, Fort Worth, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
- Otto Wagner Spital, Vienna, Austria
- France (5):
  - Hopital Henri Mondor, Créteil
  - CHU de Nice-l Archet, Nice
  - Hopital Bichat-Claude Bernard, Paris
  - Hopital Saint Louis, Paris
  - Centre Hospitalier de Tourcoing, Tourcoing
- Klinikum rechts der Isar, TUM, München, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Background] Eron JJ Jr, Lelievre JD, Kalayjian R, Slim J, Wurapa AK, Stephens JL, McDonald C, Cua E, Wilkin A, Schmied B, McKellar M, Cox S, Majeed SR, Jiang S, Cheng A, Das M, SenGupta D. Safety of elvitegravir, cobicistat, emtricitabine, and tenofovir alafenamide in HIV-1-infected adults with end-stage renal disease on chronic haemodialysis: an open-label, single-arm, multicentre, phase 3b trial. Lancet HIV. 2018 Dec 13:S2352-3018(18)30296-0. doi: 10.1016/S2352-3018(18)30296-0. Online ahead of print. PMID 30555051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe and the United States. The first participant was screened on 14 December 2015. The last study visit occurred on 15 October 2019.
Pre-assignment Details: 75 participants were screened.
Groups:
- E/C/F/TAF (GEN Phase): Participants received elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (Genvoya®, GEN) (150/150/200/10 mg) fixed-dose combination (FDC) tablet once daily with food for 96 weeks. At Week 96, participants in the United States (US) who wished to participate in the open-label (OL) rollover extension either discontinued E/C/F/TAF FDC or continued to take E/C/F/TAF FDC for up to 114 weeks.
- E/C/F/TAF to B/F/TAF (BVY OL Extension Phase): At Week 96 or the end of E/C/F/TAF visit (whichever occurred last), participants were given the option to receive open-label (OL) bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (Biktarvy®, BVY) (50/200/25 mg) FDC tablet once daily without regard to food for up to 52 weeks.
Period: GEN Phase
Arm/Group | E/C/F/TAF (GEN Phase) | E/C/F/TAF to B/F/TAF (BVY OL Extension Phase)
Started | 55 | 0
Completed | 39 | 0
Not Completed | 16 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Death | 2 | 0
Not completed — Investigator's Discretion | 4 | 0
Not completed — Non-Compliance with Study Drug | 1 | 0
Not completed — Withdrew Consent | 5 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: BVY OL Extension Phase
Arm/Group | E/C/F/TAF (GEN Phase) | E/C/F/TAF to B/F/TAF (BVY OL Extension Phase)
Started | 0 (Only US participants were eligible to roll over into the Extension Phase per the study protocol.) | 10 (Only US participants were eligible to roll over into the Extension Phase per the study protocol.)
Completed | 0 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The GEN Safety Analysis Set included all participants who received at least 1 dose of GEN.
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 45
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46
  France | 7
  Austria | 1
  Germany | 1
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 54
  ≥ 50 copies/mL | 1
Cluster Determinant 4+ (CD4+) Cell Count [Mean (Standard Deviation); unit: cells/µL] | 545 (239.2)
CD4+ Cell Count Categories [Count of Participants; unit: Participants]
  < 50 cells/µL | 0
  >= 50 to < 200 cells/µL | 0
  >= 200 to < 350 cells/µL | 12
  >= 350 to < 500 cells/µL | 14
  >= 500 cells/µL | 29
CD4 Percentage [Mean (Standard Deviation); unit: percentage of CD4 cells] | 31.5 (9.41)

OUTCOME MEASURES:

1. Primary Outcome: GEN Phase: Percentage of Participants Experiencing Treatment-Emergent Grade 3 or Higher Adverse Events Up to Week 48
Description: Treatment-emergent Adverse Events (TEAE) were defined as AEs with onset dates on or after the study drug start date and no later than 30 days after the permanent discontinuation of the E/C/F/TAF (GEN Phase) study drug or all AEs for participants still on E/C/F/TAF. It also includes the AEs that led to premature discontinuation of E/C/F/TAF study drug. Clinical events and clinically significant laboratory abnormalities were graded according to the GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities. Adverse events were graded as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), or Grade 4 (life threatening).
Time Frame: First Dose Date Up to Week 48
Population: The GEN Safety Analysis Set included participants who were enrolled and received at least 1 dose of GEN (E/C/F/TAF FDC).
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 55
percentage of participants | 32.7

2. Secondary Outcome: GEN Phase: Percentage of Participants Experiencing Treatment-Emergent Grade 3 or Higher Adverse Events Up to Week 96
Description: Treatment-emergent Adverse Events (TEAE) were defined as events that met 1 or both of the following criteria as any AEs with onset dates on or after the study drug start date and no later than 30 days after the permanent discontinuation of the E/C/F/TAF (GEN Phase) study drug for participants who did not participate in the BVY OL extension phase or the day prior to the date of the first B/F/TAF study drug dose for participants who participated in the BVY OL extension phase. It also includes the AEs that led to premature discontinuation of E/C/F/TAF study drug. Clinical events and clinically significant laboratory abnormalities were graded according to the GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities. Adverse events were graded as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), or Grade 4 (life threatening).
Time Frame: First Dose Date Up to Week 96
Population: Participants in the GEN Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 55
percentage of participants | 43.6

3. Secondary Outcome: GEN Phase: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 as Defined by the FDA Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: The GEN Full Analysis Set included participants who were enrolled and received at least 1 dose of GEN (E/C/F/TAF FDC).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 55
percentage of participants | 87.3 [75.5 to 94.7]

4. Secondary Outcome: GEN Phase: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the FDA Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the GEN Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 55
percentage of participants | 81.8 [69.1 to 90.9]

5. Secondary Outcome: GEN Phase: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96 as Defined by the FDA Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the GEN Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 55
percentage of participants | 54.5 [40.6 to 68.0]

6. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of Elvitegravir (EVG), Cobicistat (COBI), Emtricitabine (FTC), and Tenofovir (TFV)
Description: AUCtau is defined as area under the concentration versus time curve over the dosing interval (i.e., concentration of drug over time).
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose at or between Week 2 or Week 4
Population: Participants in the PK Substudy Analysis Set (participants who were enrolled into the study, participated in the intensive PK substudy, received at least 1 dose of E/C/F/TAF FDC, and had at least 1 nonmissing plasma PK concentration value for any analyte of interest) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 11
h*ng/mL
  EVG: number analyzed (Participants) | 10
  EVG | 14284.8 (7790.26)
  COBI | 10179.5 (6009.28)
  FTC | 62929.9 (30199.63)
  TFV: number analyzed (Participants) | 10
  TFV | 8715.0 (3432.16)

7. Secondary Outcome: PK Parameter: AUClast of EVG, COBI, FTC, Tenofovir Alafenamide (TAF), and TFV
Description: AUClast is defined as the area under the concentration versus time curve from time zero to the last observable concentration.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose at or between Week 2 or Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 12
h*ng/mL
  EVG | 12857.6 (7894.09)
  COBI | 9558.7 (5963.16)
  FTC | 59057.4 (31485.96)
  TAF | 231.9 (123.46)
  TFV | 7664.2 (3958.36)

8. Secondary Outcome: PK Parameter: Cmax of EVG, COBI, FTC, TAF, and TFV
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose at or between Week 2 or Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 12
ng/mL
  EVG | 1258.5 (689.57)
  COBI | 1370.4 (920.15)
  FTC | 4875.0 (1981.03)
  TAF | 246.3 (185.69)
  TFV | 442.8 (181.03)

9. Secondary Outcome: PK Parameter: Ctau of EVG, COBI, FTC, and TFV
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval. Ctau has been presented in lieu of Cmin (specified in the protocol) to align with other Gilead studies. This change has no impact on the PK analysis as Ctau and Cmin are equivalent for all analytes.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, and 24 hours postdose at or between Week 2 or Week 4
Population: Participants in the PK Substudy Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 10
ng/mL
  EVG | 174.4 (104.36)
  COBI | 28.9 (34.06)
  FTC | 1277.3 (756.60)
  TFV | 264.8 (193.98)

10. Secondary Outcome: GEN Phase: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96 Using the Missing = Failure (M = F) Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 were analyzed using the M = F approach. In this approach, all missing data was treated as HIV-1 RNA ≥ 50 copies/mL.
Time Frame: Week 96
Population: Participants in the GEN Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 55
percentage of participants | 61.8 [47.7 to 74.6]

11. Secondary Outcome: GEN Phase: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96 Using the Missing = Excluded (M = E) Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 were analyzed using the M = E approach. In this approach, all missing data was excluded in the computation of the proportions.
Time Frame: Week 96
Population: Participants in the GEN Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 34
percentage of participants | 100.0 [89.7 to 100.0]

12. Secondary Outcome: BVY OL Extension Phase: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 Using the M = E Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 were analyzed using the M = E approach. In this approach, all missing data was excluded in the computation of the proportions.
Time Frame: Week 48 of the BVY OL Extension Phase
Population: The BVY Full Analysis Set included all participants who were enrolled in the study and received at least 1 dose of BVY (B/F/TAF FDC).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF to B/F/TAF (BVY OL Extension Phase)
Number analyzed (Participants) | 10
percentage of participants | 100.0 [69.2 to 100.0]

13. Secondary Outcome: GEN Phase: Change From Baseline in Cluster Determinant 4+ (CD4+) Cell Count at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the GEN Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 28
cells/µL | -35 (218.3)

14. Secondary Outcome: BVY OL Extension Phase: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48 of the BVY OL Extension Phase
Population: Participants in the BVY Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF to B/F/TAF (BVY OL Extension Phase)
Number analyzed (Participants) | 10
cells/µL
  Baseline | 581 (146.8)
  Change from Baseline at Week 48: number analyzed (Participants) | 9
  Change from Baseline at Week 48 | -104 (120.8)

15. Secondary Outcome: GEN Phase: Change From Baseline in CD4 Percentage at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the GEN Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4 cells
Arm/Group | E/C/F/TAF (GEN Phase)
Number analyzed (Participants) | 28
percentage of CD4 cells | 2.8 (6.37)

16. Secondary Outcome: BVY OL Extension Phase: Change From Baseline in CD4 Percentage at Week 48
Time Frame: Baseline; Week 48 of the BVY OL Extension Phase
Population: Participants in the BVY Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of CD4 cells
Arm/Group | E/C/F/TAF to B/F/TAF (BVY OL Extension Phase)
Number analyzed (Participants) | 10
percentage of CD4 cells
  Baseline | 31.9 (7.37)
  Change from Baseline at Week 48: number analyzed (Participants) | 9
  Change from Baseline at Week 48 | 1.7 (4.39)

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date [maximum: 114 Weeks (GEN Phase), 52 Weeks (BVY OL Extension Phase)] plus 30 days
Description: The GEN Safety Analysis Set included all participants who received at least 1 dose of GEN.
  The BVY Safety Analysis Set included all participants who received at least 1 dose of BVY.
Arm/Group | E/C/F/TAF (GEN Phase) | E/C/F/TAF to B/F/TAF (BVY OL Extension Phase)
All-Cause Mortality (participants affected / at risk) | 3/55 | 0/10
Serious Adverse Events (participants affected / at risk) | 36/55 | 3/10
Other Adverse Events (participants affected / at risk) | 41/55 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (GEN Phase) (N=55) | E/C/F/TAF to B/F/TAF (BVY OL Extension Phase) (N=10)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardiac failure acute (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Generalised oedema (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Arteriovenous fistula site infection (Infections and infestations) | 3 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Endocarditis staphylococcal (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 4 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 0
Azotaemia (Renal and urinary disorders) | 2 | 0
End stage renal disease (Renal and urinary disorders) | 3 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Renal transplant (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Diabetic microangiopathy (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 0
Hypertensive emergency (Vascular disorders) | 2 | 1
Hypertensive urgency (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 3 | 0
Subclavian vein stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (GEN Phase) (N=55) | E/C/F/TAF to B/F/TAF (BVY OL Extension Phase) (N=10)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1
Cataract (Eye disorders) | 1 | 1
Diplopia (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Scleral hyperaemia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 13 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 3 | 0
Malaise (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 6 | 0
Peripheral swelling (General disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Electrocardiogram QT prolonged (Investigations) | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0
Headache (Nervous system disorders) | 4 | 1
Thrombosis in device (Product Issues) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Acquired phimosis (Reproductive system and breast disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 3 | 0
Superior vena cava stenosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT02600819/SAP_005.pdf
  • Study Protocol: Original (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT02600819/Prot_006.pdf
  • Study Protocol: Amendment 1 (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT02600819/Prot_007.pdf
  • Study Protocol: Amendment 2 (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT02600819/Prot_008.pdf
  • Study Protocol: Amendment 2.1 (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT02600819/Prot_009.pdf